CLINICAL TRIAL: NCT01739855
Title: Phase 2 Study of Patients Undergoing Bariatric Surgery (Laparoscopic Gastric Bypass) and Evaluation of Bone Metabolism With/Without Vitamin D/Calcium Supplementation
Brief Title: Bone Metabolism After Laparoscopic Gastric Bypass Surgery (BABS)
Acronym: BABS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christian Muschitz, Senior Consultant for Internal Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vinforce-015; Vinforce 015 (Other: Medical University Vienna)
Record Dates: First submitted 2012-11-23; First posted 2012-12-04 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Evaluation of Expected Bone Loss After Bariatric Surgery; Possible Prevention of Bone Loss After Surgery by Calcium and Vitamin D Supplementation
MeSH Terms: interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium/Vitamin D (Active Comparator): All subjects will receive calcium/vitamin D supplementation after laparoscopic bariatric gastric bypass surgery as follows:
  daily: 500 mg oral calcium (calcium carbonate) weekly: 16.000 IU oral vitamin D3 (calciferol)
  Interventions: Drug: Calciferol, calcium carbonate
- No Calcium/Vitamin D (No Intervention): All subjects will not receive calcium/vitamin D supplementation after laparoscopic bariatric gastric bypass surgery.

INTERVENTIONS:
Drug: Calciferol, calcium carbonate
  Arms: Calcium/Vitamin D

SUMMARY:
Bariatric surgery leads to rapid weight loss in female and male patients. Less data are available about its impact on bone metabolism.

The aim of this study is the investigation of changes in bone mineral density,bone histomorphometric changes, serum bone turnover markers and changes in body fat and muscle composition in patients after laparoscopic gastric bypass surgery.

DETAILED DESCRIPTION:
Obese female and male adult patients eligible for laparoscopic gastric bypass surgery according to the national Austrian guidelines will be included in this study upon request and after patient approval.

Baseline data collection and quarterly follow up visits are planned to investigate the changes in bone mineral density and body composition measured by dual energy X-ray absorptiometry as well as the evaluation of serum bone turnover markers of bone formation and resorption.

After surgery subjects will be randomized into two groups:

Daily oral calcium (500mg) and weekly vitamin D3 supplementation (16.000 IU calciferol)or no supplementation of calcium and calciferol.

A sub-study (approximately 15% of study population) with transiliac bone biopsies will also be performed to investigate histomorphometric and histologic changes in bone (biopsy baseline and after 24 months).

The planned duration of the study is 24 months for each subject. Serum bone turnover markers will be collected every 3 months, dual energy X-ray absorptiometry measurements will be performed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* body mass index >35
* female and male patients
* age 18 - 65 years
* eligible for laparoscopic gastric bypass surgery according to the Austrian national guidelines

Exclusion Criteria:

* any history of malignancy except basalioma
* any prior antiresorptive treatment
* any prior calcium or vitamin D supplementation
* any secondary disease affecting bone metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of bone mineral density changes in obese patients after laparoscopic bariatric surgery | Evaluation every 6 months for 24 months
  Dual energy X-ray absorptiometry (DXA) measurements of bone mineral density at lumbar spine, hip, calcaneus and total body will be performed at baseline and every six months for a period of 24 months.
  Differences will be evaluated on the outcome with/without daily calcium (500mg) and weekly vitamin D (16.000 IU calciferol) supplementation

SECONDARY OUTCOMES:
Evaluation of changes of serum bone turnover markers in obese patients after laparoscopic bariatric surgery | Evaluation every 3 months for 24 months
  Fasting serum markers of bone formation and bone resorption will be evaluated:
  Calcium, 25-OH-vitamin D3, intact parathyroid hormone, beta-crosslaps, type-1-procollagen, bone specific alkaline phosphatase, osteocalcin, sclerostin, osteoprotegerin, cathepsin-K, fibroblast factor 23, lipoprotein A, dickkopf 1 Differences will be evaluated on the outcome with/without daily calcium (500mg) and weekly vitamin D (16.000 IU calciferol) supplementation

OTHER OUTCOMES:
Evaluation of histomorphometric and histologic changes in obese patients after laparoscopic bariatric surgery | baseline and after 24 months
  Transiliac bone biopsies will be performed in a approximately 15% of patients at baseline and after 24 months.
  The following parameters will be measured: bone volume (BV/TV), bone surface (BS/BV), osteoblast surface (OS/BS), trabecular number (TbN), trabecular thickness (TbTh, trabecular separation (Tb.sp), mineralized surface (MS/BS), mineral apposition rate (MAR) Differences will be evaluated on the outcome with/without daily calcium (500mg) and weekly vitamin D (16.000 IU colecalciferol) supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Muschitz, M.D., Principal Investigator — Medical University Vienna - Austria
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Muschitz C, Kocijan R, Haschka J, Zendeli A, Pirker T, Geiger C, Muller A, Tschinder B, Kocijan A, Marterer C, Nia A, Muschitz GK, Resch H, Pietschmann P. The Impact of Vitamin D, Calcium, Protein Supplementation, and Physical Exercise on Bone Metabolism After Bariatric Surgery: The BABS Study. J Bone Miner Res. 2016 Mar;31(3):672-82. doi: 10.1002/jbmr.2707. Epub 2015 Sep 30. PMID 26350034